CLINICAL TRIAL: NCT00006059
Title: Genetic Study of Familial Epilepsy
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Columbia University (Other)
Other Study IDs: NCRR-M01RR00645-2635; CPMC-IRB-4465
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Epilepsy
Keywords: epilepsy; neurologic and psychiatric disorders; rare disease; seizures
MeSH Terms: conditions — Epilepsy; Neurologic Manifestations; Mental Disorders; Rare Diseases; Seizures

SUMMARY:
OBJECTIVES:

I. Determine the chromosomal regions that contain genes that raise the risk of epilepsy in families by performing genetic linkage analysis of idiopathic/cryptogenic epilepsy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Family histories are obtained, then the patients undergo an interview, a neurological examination, and EEG. Blood specimens are also collected.

Linkage analysis is performed on specimens and analysis of shared marker alleles are used to identify genomic regions likely or unlikely to contain the epilepsy genes. Genotypes in family members are determined at microsatellite markers throughout the genome. Markers tested include chromosomes linked to human epilepsy syndromes (6p, 8p, 8q, 20q, 21q) and chromosome 3 (similar to mouse "epilepsy" genes). Linkage to markers on chromosome 10q are also tested.

Patients do not receive the results of the testing and the results do not influence the type and duration of any treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Male or female members of families with at least 1 close relative pair (sibling, half sibling, avuncular, grandparent-grandchild, or first cousin) affected with idiopathic/cryptogenic epilepsy that developed before age 25

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 898
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Ottman, Study Chair — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States